CLINICAL TRIAL: NCT00412724
Title: Development and Validation of the Food Acceptability Questionnaire
Status: Completed | Type: Observational
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: FAQ
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: diet; acceptability; palatability; food; questionnaire; Food habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Food Acceptability Questionnaire (FAQ) is a self-report measure of palatability, ease of preparation, satisfaction, and perceived benefits and adverse effects related to a prescribed or self-selected diet. This study intends to develop a reliable and valid food acceptability questionnaire for use in clinical studies in which dietary interventions are administered.

DETAILED DESCRIPTION:
Two hundred adult participants who follow a therapeutic diet will be recruited from the Washington DC area. Participants will be asked to rate their impression on the foods that they were eating in the past two weeks. Fifty participants will be chosen at random and asked to complete the questionnaire a second time, three weeks later, to assess reliability. Ratings will be used to assess the validity and reliability of the Food Acceptability Questionnaire (FAQ).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be older than 18 years and follow any kind of therapeutic diet.

Exclusion Criteria:

* Those who have difficulty eating by themselves will be excluded. No vulnerable subjects will be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women following a theraputic diet for at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Ahlgren SS, Shultz JA, Massey LK, Hicks BC, Wysham C. Development of a preliminary diabetes dietary satisfaction and outcomes measure for patients with type 2 diabetes. Qual Life Res. 2004 May;13(4):819-32. doi: 10.1023/B:QURE.0000021694.59992.a1. PMID 15129892
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] White MA, Whisenhunt BL, Williamson DA, Greenway FL, Netemeyer RG. Development and validation of the food-craving inventory. Obes Res. 2002 Feb;10(2):107-14. doi: 10.1038/oby.2002.17. PMID 11836456
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681